CLINICAL TRIAL: NCT03773055
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Parallel Group Trial to Investigate the Proof of Concept of NPC-06 in Patients With Neuropathic Pain in Cancer
Brief Title: Phase II Clinical Trial of NPC-06 in Patients With Neuropathic Pain in Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NPC-06-4
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-08

CONDITIONS: Neuropathic Pain in Cancer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NPC-06 (High dosage) (Active Comparator): 18 mg (iv) in Day 1 as an induction dosage and 9 mg (iv) in Day 2 - 7 as a maintenance dosage
  Interventions: Drug: NPC-06
- NPC-06 (Low dosage) (Active Comparator): 15 mg (iv) in Day 1 as an induction dosage and 6 mg (iv) in Day 2 - 7 as a maintenance dosage
  Interventions: Drug: NPC-06
- Placebo (Placebo Comparator): Saline will be administered intravenously
  Interventions: Drug: NPC-06

INTERVENTIONS:
Drug: NPC-06 — Patients will receive once a day for 7 days.

SUMMARY:
The purpose of this trial is to investigate the efficiency of pain relief and the safety of NPC-06 for the neuropathic pain associated with cancer, in addition to explore the effective concentration of NPC-06.

DETAILED DESCRIPTION:
The eligible patients will be randomized into three groups, and will receive NPC-06 (high dose), NPC-06 (low dose) or placebo once a day for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. 16 years old or greater at the time of informed consent
2. Both genders
3. Patients who can admit to hospital for all assessment duration from first administration until the next day of final administration. (including the hospitalized patient )
4. Patients who are diagnosed and informed as cancer (including sarcoma, lymphoma and multiple myeloma)
5. Patients who are diagnosed as neuropathic pain by neurological examination and imaging findings
6. Patients who NRS score of average persistent pain is higher than 4, even they were treated with level 3 of WHO three-step analgesic ladder at the observation period.
7. Patients who NRS score at the time of first administration and NRS score of persistent pain in the past 24 hours are higher than 4.
8. Patients who average number of daily rescue medication use during observation period is less than 6.
9. Patients who are predicted to survive longer than 3 month.
10. Patients who ECOG Performance Status (PS) score is 0 to 3.
11. Patients who (or whose legally acceptable representative if the patient is underage) provide a written consent at their own will with a full understanding after receiving a sufficient explanation on participation in the study

Exclusion Criteria:

1. Patients who can not evaluate NRS by themselves.
2. Patients who have leukemia as a complication.
3. Patients who have a primary brain neoplasm or a metastatic brain neoplasm as a complication.
4. Patients who have epilepsy, serious psychiatric or neurological disease ( i. e. dementia, Parkinson disease or schizophrenic disorder) or consciousness disturbance as a complication.
5. Patients who have primary trigeminal neuralgia, diabetic neuropathy, post herpetic neuralgia or acute herpes zoster pain as a complication.
6. Patients who has other serious pain which affect the evaluation of neuropathic pain in cancer.
7. Patients who have sinus bradycardia or serious disturbance of conduction system.
8. Patients who have history of hypersensitivity against hydantoin compound.
9. Patients who are administrated tadalafil (for pulmonary hypertension), rilpivirine, asunaprevir, daclatasvir, vaniprevir, macitentan or sofosbuvir.
10. Patients who are administrated methadone.
11. Patients who have complications such as serious heart disease, hepatic function disorder or renal function disorder which severity are considered by investigator as grade 3 or more severe with reference to ''Concerning classification criteria for seriousness of adverse drug reactions of medical agents'' (except cancer).
12. Patients who received surgical treatment or internal radiation therapy in past three month before the first day of pre observation period.
13. Patients who are treated nerve block, radiation therapy, spinal cord stimulation or surgical treatment for the part of neuropathic pain in past one month before the first day of pre observation period.
14. Patients who change the usage or dosage of medication for cancer as primal disease in the past two week before the first day of the pre observation period, or patients who are predicted not to continue the treatment without change in the medication while this clinical trial.
15. Patients who are administrating with fosphenytoin, phenytoin or ethotoin or have taken these drugs as medication for neuropathic pain.
16. Patients who have participated in other clinical trial and have taken a trial drug in past three month before the first day of pre observation period.
17. Female patients who are pregnant or lactating or who may be pregnancy in the period of the clinical trial.
18. Patients who can not agree to prevent contraception appropriately following the direction of the Investigator or the sub-investigator.
19. Any other patients who are considered by the investigator as unsuitable for participation in the trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Improvement of Numeric Rating Scale (NRS) score within 2 hours after administration | Pre-administration, 30, 60, 90 and 120 minutes post-administration
  Average change (slope) of NRS score

SECONDARY OUTCOMES:
Other improvements of NRS score | Pre-dose, Days 1,2,3,4,5,6,7,8,9,10,11,12,13
  Change of NRS score, Change of NRS score of persistent pain, Change of maximum pain, at the time of evaluation compared to baseline
Time to event | 2 hours after initial administration to Day 7
  Time to event analysis of analgesic effect
Improvement of Neuropathic Pain Symptom Inventory (NPSI) score | Pre-dose, Days 1,2,3,4,5,6,7,8,9,10,11,12,13
  Change of NPSI score compared to baseline
Rescue medication use | Day 1 to Day 13
  Number of times of rescue medication use
Effective concentration | Day 0 to Day 13
  Blood phenytoin concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Keio Hospital, Shinjuku-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No